CLINICAL TRIAL: NCT04635254
Title: Effects of Halophyte-based Cream Skin Application in a Human Experimental Model of Pain and Itch
Brief Title: The Effect of Halophyte-based Cream on Pain and Itch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Rocco Giordano, Principal Investigator, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20200072
Record Dates: First submitted 2020-10-28; First posted 2020-11-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Pain, Acute; Itch
MeSH Terms: conditions — Acute Pain; Pruritus | interventions — Tumor Protein, Translationally-Controlled 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Halophites-based cream 24 hours (Active Comparator): A 2 gram amount of Halophites-based cream will be applied under occlusion (TegaDerm tape) in a 4x4 cm squared area.
  Interventions: Other: Halophites-based cream 24 hours; Other: Vehicle cream 24 hours; Other: Histamine 1%; Other: Cowhage
- Halophites-based cream 48 hours (Active Comparator): A 2 gram amount of Halophites-based cream will be applied under occlusion (TegaDerm tape) in a 4x4 cm squared area.
  Interventions: Other: Halophites-based cream 48 hours; Other: Vehicle cream 48 hours; Other: Histamine 1%; Other: Cowhage

INTERVENTIONS:
Other: Halophites-based cream 24 hours — The concentration of active aqueous extract will be in the range of 2% to 30% (v/v) by cold emulsification. A 2 gram amount of Halophytes-based cream will be applied under occlusion (TegaDerm tape) in a 4x4 cm squared area.
  Arms: Halophites-based cream 24 hours
Other: Halophites-based cream 48 hours — The concentration of active aqueous extract will be in the range of 2% to 30% (v/v) by cold emulsification. A 2 gram amount of Halophytes-based cream will be applied under occlusion (TegaDerm tape) in a 4x4 cm squared area.
  Arms: Halophites-based cream 48 hours
Other: Vehicle cream 24 hours — A 2 gram amount of vehicle cream will be applied under occlusion (TegaDerm tape) in a 4x4 cm squared area.
  Arms: Halophites-based cream 24 hours
Other: Vehicle cream 48 hours — A 2 gram amount of vehicle cream will be applied under occlusion (TegaDerm tape) in a 4x4 cm squared area.
  Arms: Halophites-based cream 48 hours
Other: Histamine 1% — To deliver histamine, standard allergy skin prick test (SPT) lancets are applied. The lancets have a 1 mm shouldered tip adapt to introduce a small amount of test substance extremely locally and approximately at the dermo-epidermal junction.
Other: Cowhage — The insertion of cowhage spicule(s) rapidly and consistently produces itch with no or very little flare reaction. This insertion is conducted by forceps using a stereo-microscope, and 30-35 spicules are gently rubbed into a 1 cm diameter skin area.

SUMMARY:
In this study the investigators wish to investigate whether halophyte-based cream applied to the skin can reduce itch applied by means of small needles from the plant mucuna pruriens (also called cowhage) or by histamine (an itch-evoking substance formed in the human body). Further, the investigators wishes to investigate whether long-term application of halophyte-based cream has a pain-relieving effect on heat/cold and pinprick stimulations.

DETAILED DESCRIPTION:
Salt-tolerant plants (also called halophytes) can grow in saline soil or directly in salt water (e.g. along coasts). For centuries, these plants have been used in folk medicine, and among other things they are believed to have pain-relieving and anti-inflammatory effect.

Even though experiments have already investigated halophytes as a pain relieving substance, the mechanisms in relation to pain and/or itch are still unknown. Therefore, the investigators wish to investigate whether halophyte-based cream applied to the skin can reduce itch applied by means of small needles from the plant mucuna pruriens (also called cowhage) or by histamine (an itch-evoking substance formed in the human body). Further, the investigators wishes to investigate whether long-term application of halophyte-based cream has a pain-relieving effect on heat/cold and pinprick stimulations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids or other drugs
* Previous or current neurologic, musculoskeletal or mental illnesses that may affect the results (e.g. neuropathy, muscular pain in the upper extremities, etc.)
* Lack of ability to cooperate
* Current use of medications that may affect the trial such as antihistamine medications or pain killers
* Skin diseases
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical trials)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Superficial blood perfusion | Day 0
  Superficial blood perfusion is measured by a Speckle contrast imager (FLPI, Moor Instruments, England).
Superficial blood perfusion | 24 hours after cream application
  Superficial blood perfusion is measured by a Speckle contrast imager (FLPI, Moor Instruments, England).
Superficial blood perfusion | 48 hours after cream application
  Superficial blood perfusion is measured by a Speckle contrast imager (FLPI, Moor Instruments, England).
Itch intensity | Day 0
  The subject will rate the itch sensation on a 100 millimeter Visual Analog Scale from 0 to 100., where 0"indicates no itch and "100" worst itch imaginable
Itch intensity | 24 hours after cream application
  The subject will rate the itch sensation on a 100 millimeter Visual Analog Scale from 0 to 100., where 0"indicates no itch and "100" worst itch imaginable
Itch intensity | 48 hours after cream application
  The subject will rate the itch sensation on a 100 millimeter Visual Analog Scale from 0 to 100., where 0"indicates no itch and "100" worst itch imaginable
Pain intensity | Day 0
  The subject will rate the pain sensation on a 100 millimeter Visual Analog Scale from 0 to 100., where 0"indicates no pain and "100" worst pain imaginable
Pain intensity | 24 hours after cream application
  The subject will rate the pain sensation on a 100 millimeter Visual Analog Scale from 0 to 100., where 0"indicates no pain and "100" worst pain imaginable
Pain intensity | 48 hours after cream application
  The subject will rate the pain sensation on a 100 millimeter Visual Analog Scale from 0 to 100., where 0"indicates no pain and "100" worst pain imaginable
Measuring Alloknesis | Day 0
  Alloknesis is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).
Measuring Alloknesis | 24 hours after cream application
  Alloknesis is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).
Measuring Alloknesis | 48 hours after cream application
  Alloknesis is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).
Trans-epidermal Water Loss (TEWL) | Day 0
  TEWL is a non-invasive and pain free measuring technique in which a 2x2 cm hollow probe with two small humidity gauges and two thermometers is placed lightly on the skin for 10-25 seconds. These collectively establish a precise humidity gradient in a 2 cm vicinity of the skin, representative for the point-loss of water though the epidermis.
Trans-epidermal Water Loss (TEWL) | 24 hours after cream application
  TEWL is a non-invasive and pain free measuring technique in which a 2x2 cm hollow probe with two small humidity gauges and two thermometers is placed lightly on the skin for 10-25 seconds. These collectively establish a precise humidity gradient in a 2 cm vicinity of the skin, representative for the point-loss of water though the epidermis.
Trans-epidermal Water Loss (TEWL) | 48 hours after cream application
  TEWL is a non-invasive and pain free measuring technique in which a 2x2 cm hollow probe with two small humidity gauges and two thermometers is placed lightly on the skin for 10-25 seconds. These collectively establish a precise humidity gradient in a 2 cm vicinity of the skin, representative for the point-loss of water though the epidermis.

SECONDARY OUTCOMES:
Measurement of Warm Detection Thresholds (WDT) | Day 0
  The tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. During the first 8 seconds, the temperature raises 1°C per second from a starting temperature of 32°C until the subject perceives a temperature change (warm sensation) and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 52°C will be used.
Measurement of Warm Detection Thresholds (WDT) | 24 hours after cream application
  The tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. During the first 8 seconds, the temperature raises 1°C per second from a starting temperature of 32°C until the subject perceives a temperature change (warm sensation) and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 52°C will be used.
Measurement of Warm Detection Thresholds (WDT) | 48 hours after cream application
  The tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. During the first 8 seconds, the temperature raises 1°C per second from a starting temperature of 32°C until the subject perceives a temperature change (warm sensation) and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 52°C will be used.
Measurement of Cold Detection Thresholds (CDT) | Day 0
  The tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. During the first 8 seconds, the temperature decreases 1°C per second from a starting temperature of 32°C until the subject perceives a temperature change (cold sensation) and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 0°C will be used.
Measurement of Cold Detection Thresholds (CDT) | 24 hours after cream application
  The tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. During the first 8 seconds, the temperature decreases 1°C per second from a starting temperature of 32°C until the subject perceives a temperature change (cold sensation) and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 0°C will be used.
Measurement of Cold Detection Thresholds (CDT) | 48 hours after cream application
  The tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. During the first 8 seconds, the temperature decreases 1°C per second from a starting temperature of 32°C until the subject perceives a temperature change (cold sensation) and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 0°C will be used.
Measurement of Heat Pain Thresholds (HPT) | Day 0
  The tests for thermal sensation will all be performed using the same PATHWAY ATS thermal sensory testing device as above. The stimulations are again applied on the treated/placebo areas. During the first 8 seconds, the temperature raises 1°C per second from a starting temperature of 32°C until the subject detects a painful sensation and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 52°C will be used.
Measurement of Heat Pain Thresholds (HPT) | 24 hours after cream application
  The tests for thermal sensation will all be performed using the same PATHWAY ATS thermal sensory testing device as above. The stimulations are again applied on the treated/placebo areas. During the first 8 seconds, the temperature raises 1°C per second from a starting temperature of 32°C until the subject detects a painful sensation and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 52°C will be used.
Measurement of Heat Pain Thresholds (HPT) | 48 hours after cream application
  The tests for thermal sensation will all be performed using the same PATHWAY ATS thermal sensory testing device as above. The stimulations are again applied on the treated/placebo areas. During the first 8 seconds, the temperature raises 1°C per second from a starting temperature of 32°C until the subject detects a painful sensation and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 52°C will be used.
Measurement of Cold Pain Thresholds (CPT) | Day 0
  The tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. During the first 8 seconds, the temperature decreases 1°C per second from a starting temperature of 32°C until the subject detects a painful sensation and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 0°C will be used.
Measurement of Cold Pain Thresholds (CPT) | 24 hours after cream application
  The tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. During the first 8 seconds, the temperature decreases 1°C per second from a starting temperature of 32°C until the subject detects a painful sensation and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 0°C will be used.
Measurement of Cold Pain Thresholds (CPT) | 48 hours after cream application
  The tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. During the first 8 seconds, the temperature decreases 1°C per second from a starting temperature of 32°C until the subject detects a painful sensation and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 0°C will be used.
Measurement of Pain to Supra-threshold Heat Stimuli: | Day 0
  Again, the tests will be performed by using the PATHWAY ATS thermal sensory testing device. The subjects will have to rate the pain to three suprathreshold heat pain stimuli (starting and ending at 34°C with an increase and decrease of 5°C and 4 s plateau at 50°C) applied on the treated/placebo areas .
Measurement of Pain to Supra-threshold Heat Stimuli: | 24 hours after cream application
  Again, the tests will be performed by using the PATHWAY ATS thermal sensory testing device. The subjects will have to rate the pain to three suprathreshold heat pain stimuli (starting and ending at 34°C with an increase and decrease of 5°C and 4 s plateau at 50°C) applied on the treated/placebo areas .
Measurement of Pain to Supra-threshold Heat Stimuli: | 48 hours after cream application
  Again, the tests will be performed by using the PATHWAY ATS thermal sensory testing device. The subjects will have to rate the pain to three suprathreshold heat pain stimuli (starting and ending at 34°C with an increase and decrease of 5°C and 4 s plateau at 50°C) applied on the treated/placebo areas .
Measurement of Mechanical Pain Thresholds (MPT) | Day 0
  This test is performed using a pin-prick set (Aalborg University, Aalborg). The set consists of 8 needles each having a diameter of 0.6 mm and different force applications: 0.8, 1.6, 3.2, 6.4, 12.8, 25.6, 50.1 and 60.0 g. Starting with the lightest, each stimulator is applied at a rate of 2 s on, 2 s off in an ascending order until the first perception of sharpness is reached. The final threshold is the geometric mean of five series of ascending and descending stimuli.
Measurement of Mechanical Pain Thresholds (MPT) | 24 hours after cream application
  This test is performed using a pin-prick set (Aalborg University, Aalborg). The set consists of 8 needles each having a diameter of 0.6 mm and different force applications: 0.8, 1.6, 3.2, 6.4, 12.8, 25.6, 50.1 and 60.0 g. Starting with the lightest, each stimulator is applied at a rate of 2 s on, 2 s off in an ascending order until the first perception of sharpness is reached. The final threshold is the geometric mean of five series of ascending and descending stimuli.
Measurement of Mechanical Pain Thresholds (MPT) | 48 hours after cream application
  This test is performed using a pin-prick set (Aalborg University, Aalborg). The set consists of 8 needles each having a diameter of 0.6 mm and different force applications: 0.8, 1.6, 3.2, 6.4, 12.8, 25.6, 50.1 and 60.0 g. Starting with the lightest, each stimulator is applied at a rate of 2 s on, 2 s off in an ascending order until the first perception of sharpness is reached. The final threshold is the geometric mean of five series of ascending and descending stimuli.
Measurement of Mechanical Pain Sensitivity (MPS) | Day 0
  This test is performed using the same pin-prick set as for the MPT test. Starting with the lightest, each stimulator is applied at a rate of 2 s on, 2 s off in an ascending order, and the subject will be asked to give a pain rating for each stimulus on a scale from 0-10 (where 0 indicates ''no pain'', and 10 indicates the ''worst imaginable pain''). This procedure will be repeated twice.
Measurement of Mechanical Pain Sensitivity (MPS) | 24 hours after cream application
  This test is performed using the same pin-prick set as for the MPT test. Starting with the lightest, each stimulator is applied at a rate of 2 s on, 2 s off in an ascending order, and the subject will be asked to give a pain rating for each stimulus on a scale from 0-10 (where 0 indicates ''no pain'', and 10 indicates the ''worst imaginable pain''). This procedure will be repeated twice.
Measurement of Mechanical Pain Sensitivity (MPS) | 48 hours after cream application
  This test is performed using the same pin-prick set as for the MPT test. Starting with the lightest, each stimulator is applied at a rate of 2 s on, 2 s off in an ascending order, and the subject will be asked to give a pain rating for each stimulus on a scale from 0-10 (where 0 indicates ''no pain'', and 10 indicates the ''worst imaginable pain''). This procedure will be repeated twice.

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, Denmark